CLINICAL TRIAL: NCT02103543
Title: A Randomized Trial in Patients With Lumbar Spinal Stenosis, Comparing the Order of Treatment With Epidural Corticosteroid Injections and Physical Therapy
Brief Title: Comparison of the Order of Treatment in Lumbar Spinal Stenosis
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of recruitment
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Hassan Monfared MD, Assistant Professor, Program Director, Emory University
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB00061868
Record Dates: First submitted 2014-03-27; First posted 2014-04-04 (Estimated); Last update posted 2017-02-23 (Actual); Status verified 2017-02

CONDITIONS: Lumbar Spinal Stenosis
MeSH Terms: conditions — Spinal Stenosis | interventions — Physical Therapy Modalities

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Physical Therapy first (Active Comparator): patients will undergo physical therapy 3-4 sessions followed by lumbar interlaminar epidural steroid injection
  Interventions: Other: physical therapy; Procedure: lumbar interlaminar epidural steroid injection; Drug: epidural steroid injection
- lumbar epidural steroid first (Active Comparator): lumbar interlaminar epidural steroid injection followed by patients will undergo physical therapy 3-4 sessions
  Interventions: Other: physical therapy; Procedure: lumbar interlaminar epidural steroid injection; Drug: epidural steroid injection

INTERVENTIONS:
Other: physical therapy — physical therapy consisting of core strengthening, low back stretching and range of motion 3 sessions
Procedure: lumbar interlaminar epidural steroid injection — single lumbar interlaminar epidural steroid injection
Drug: epidural steroid injection — Dexamethasone 10mg or Depomedrol 40mg, together with Bupivacaine 0.25% (for 3-5mL total injectate volume)

SUMMARY:
Patients with back pain with spinal stenosis of the lower back will be asked to volunteer for this research study. These patients don't need immediate surgery for this problem. Treatment of this kind of back pain with spinal stenosis usually includes physical therapy exercises and steroid injections. Both treatments are usually helpful in patients with back pain with spinal stenosis. However, physicians and other healthcare providers don't know which treatment is better to give first. The purpose of this research is to answer that question. Patients enrolled in this study will receive both treatments: physical therapy (PT) and a steroid injection ("shot"). However, patients may get the shot first followed by PT, or they may have PT first, followed by the shot. Their time in this study will last up to 6 months, and there will be five outcome measurements (via visits or telephone). All study visits will take place at the Atlanta VA Medical Center (Atlanta VA). Investigators hope to enroll about 120 subjects from the Atlanta VA. Enrolled patients will be randomized using a randomization computer program.

ELIGIBILITY:
Inclusion Criteria: chronic low back pain (at least 3 months in duration), a Visual Analogue Scale (VAS) greater than 30 (on a 100 point scale), between the ages of 18 to 80 years, either without radiating leg pain (below the knees) or with low back and/or buttock pain greater than leg pain (in which case the VAS for leg pain must be 20 or less), ability to read English and complete the assessment instruments, and diagnosis of lumbar spinal stenosis by a board certified radiologist or a board certified physiatrist either by magnetic resonance imaging (MRI) or computed-tomography (CT) that has previously been done as part of a normal course of patients medical treatment. All underlying etiology or diagnoses that are the source for lumbar spinal stenosis will be recorded (e.g. spondylolisthesis, herniated or degenerative discs, spondylosis).

-

Exclusion Criteria:

* history of lumbar surgery, acute disc herniation as reported on a radiologic imaging report, acute or severe chronic illness that are unstable, cognitive impairment which prevents the patient from providing accurate data or giving informed consent, neurological conditions (e.g. stroke, Parkinson's, brain injury), lower extremity amputees, fibromyalgia or chronic generalized pain, unstable opioid use or any signs or evidence of alcohol dependence or illicit drug use (as determined by screening questionnaire), clinical suspicion of facet joint-originating back pain or a positive response to prior facet joint block, lumbar epidural steroid injections within the last 6 months, uncontrolled psychiatric disorders, serious concomitant medical illness (e.g. acute heart failure, acute renal failure) or severe pain that may impair patient's ability to participate in physical therapy exercises or pain that is deemed so severe such that withholding of an ESI until after completion of the PT exercises is seen as causing unreasonable suffering to the patient, and conditions that would prevent the patient from undergoing fluoroscopy (e.g. pregnancy).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-01 (Estimated); Primary Completion 2017-01 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Oswestry disability Index | 1 year
  measurements will be done at baseline, week 4 (1-2 weeks after intervention), 6 months, and at 1 year

SECONDARY OUTCOMES:
visual analog scale | 1 year
  measurements will be done at baseline, week 4 (1-2 weeks after intervention), 6 months, and at 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Hassan Monfared, MD, Study Director — Emory University
Locations (1):
- Atlanta Veterans Affairs Medical Center, Decatur, Georgia, United States